CLINICAL TRIAL: NCT03010514
Title: A Chinese Registry to Determine the Genetic Risk Factors and Serumal Biomarkers for Thoracic Aortic Aneurysm/Dissection
Brief Title: A Registry Study on Genetics and Biomarkers of Thoracic Aortic Aneurysm/Dissection
Acronym: ARSGBTAAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: BeijingIHLBVD2016017
Record Dates: First submitted 2016-12-21; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Aortic Aneurysm, Thoracic; Aneurysm, Dissecting
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — If a blood specimen is obtained, it will be separated and stored at -80 ℃ as plasma, viable cells, and extracted DNA. If a saliva specimen is obtained, it is stored for DNA.
  If a tissue specimen is obtained, it will be cut into small pieces and stored at liquid nitrogen.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- case
- control

SUMMARY:
This is a national registry study to determine genetic risk factor and serial biomarkers of thoracic aortic aneurysm/dissection

ELIGIBILITY:
Case Inclusion Criteria:

1. Subject who was diagnosed as thoracic aortic aneurysm/dissection by CT angiography, interventional angiography or vascular ultrasound;
2. Age is less than 80 years old;
3. male and non pregnancy female;
4. Subject understands study requirements aand agrees to sign an informed consent form prior to any study procedures.

Case Exclusion Criteria:

Subject has one of the following:

1. Pseudoaneurysm;
2. Previous infection or trauma in the damaged part of aorta;
3. Pregnancy female;
4. Participate in other clinical trials in the last 1 months.

Control Inclusion Criteria:

1. Age and gender are matched with cases;
2. No aortic disease was detected by outpatient ultrasound;
3. No family history of cardiovascular disease;
4. Normal biochemical indicators;

Criteria for culling, shedding and suspension testing:

1. Culling: Unqualified cases and controls. Data of culled subjects can not be used for statistical analysis;
2. Shedding: Subject that self withdrawal, loss to follow-up, or quitted by doctors; Reasons for shedding should be indicated for each shed subject.
3. Suspension: a) The researchers found significant safety problems or wrong study design; b) Researchers cannot continue clinical research due to funding or management reasons; c) Director ends the study. When suspension happens, all the CRF table should be reserved for future reference.

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: case group consists of patients who was diagnosed as thoracic aortic aneurysm/dissection; control group is general population without aortic aneurysm/dissection
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-10; Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Age for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Gender for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Height for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Weight for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Contact information for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Past Medical History including disease history, surgical history, and family medical history | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Lifestyle including smoking history and drinking, specify how many years smoking or drinking lasted and detail quantity per day | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Exon sequencing data of each participant | Sequencing will be carried out in an average of 3 months after sample recruiting
Serum biomarker screening data of each participant | Screening will be carried out in an average of 3 months after sample recruiting
The location of Aneurysm/Dissection | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
The size of Aneurysm/Dissection | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：blood lipid | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：blood glucose | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：uric acid | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：urea | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：creatinine | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：C reactive protein | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：d dime | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Drug treatment | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Surgery type | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Prognosis information: all-cause death | These data is collected during follow-up visit at 3/6/12 months after discharge
Prognosis information: whether recidivation happened | These data is collected during follow-up visit at 3/6/12 months after discharge
Prognosis information including: whether other related disease happened | These data is collected during follow-up visit at 3/6/12 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jie Du, PHD, Study Director — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fang G, Tian Y, Huang S, Zhang X, Liu Y, Li Y, Du J, Gao S. KLF15 maintains contractile phenotype of vascular smooth muscle cells and prevents thoracic aortic dissection by interacting with MRTFB. J Biol Chem. 2024 May;300(5):107260. doi: 10.1016/j.jbc.2024.107260. Epub 2024 Apr 4. PMID 38582447